CLINICAL TRIAL: NCT04316078
Title: A Novel Patient Engagement Platform Used to Improve Understanding, Treatment Compliance and Quality of Care Among Patients With Gastrointestinal Malignancies
Brief Title: A Novel Patient Engagement Platform Among Patients With Gastrointestinal Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHEBA-19-6013-YL-CTIL
Record Dates: First submitted 2020-02-23; First posted 2020-03-20 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2020-03

CONDITIONS: Colon Cancer; Gastric Cancer; Pancreas Cancer; Rectal Cancer; Cholangiocarcinoma; Small Bowel Cancer; Esophageal Cancer
Keywords: patient reported outcome; quality of life; personalized videos
MeSH Terms: conditions — Colonic Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Cholangiocarcinoma; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized control study (2:1 allocation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- personalized engagement platform (Experimental): Patients registered into personalized engagement platform (PEP) will receive personalized educational videos (PEV) according to disease, treatment protocol and side effects.
  Interventions: Other: patient engagement platform
- control group (No Intervention): The control group will not be registered to the PEP nor receive any PEVs.

INTERVENTIONS:
Other: patient engagement platform — 1. Allows patients to receive the action plan as educational videos on demand.
  2. Allows patients to report side effects and quality of life via questionnaires and receive immediate targeted education based on the predefined action plan.
  Arms: personalized engagement platform

SUMMARY:
A randomized control trial to evaluate the feasibility of implementing a patient educational platform (PEP) for patients with gastrointestinal malignancies undergoing active chemotherapy treatment.

DETAILED DESCRIPTION:
Patients will be randomized in a 2:1 ratio.

Patients in the experimental arm will receive automatically generated personalized educational videos (PEV) and questionnaires regarding side effects and quality of life (QOL) to either their cell phone or email. The videos will be personalized to each patient based on their demographics, specific medical instructions and treatment plan. Data collected regarding side effects and QOL in the experimental arm will be used in order to facilitate real time intervention through real time provider alert system.

A link to the first PEV will be sent before the first chemotherapy cycle, addressing the diagnosis and type of malignancy, chemotherapy protocol, common side effects and their management. Side effects questionnaire will be sent every week while QOL questionnaire will be sent every 6 weeks.

Patients will be followed from recruitment through three weeks after completion of the planned treatment protocol. If treatment is discontinued prior to completion of the protocol, follow-up will end three weeks after the last administered treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a newly diagnosed gastrointestinal malignancy, treated at the outpatient clinic of the Institute of Oncology at the Sheba Medical Center
2. Individuals planned to receive one of the following cytotoxic chemotherapy protocols:

   1. FOLFOX - a combination of 5-fluoruracil, leucovorin and oxaliplatin.
   2. FOLFOIRI - a combination of 5-fluoruracil, leucovorin and irinotecan.
   3. FOLFIRINOX - a combination of 5-fluoruracil, leucovorin, oxaliplatin and irinotecan.
   4. De Gramont - 5-fluoruracil and leucovorin.
3. Ability to read and comprehend Hebrew language text.
4. Ability to see computer or cell phone screen (i.e., no visual impairment).

Exclusion Criteria:

1. Eastern Conference Oncology Group (ECOG) performance status greater than 2.
2. Cognitive deficits that would preclude understanding of consent form and/or questionnaires.
3. Inability to read and comprehend Hebrew language text.
4. Current participation in a therapeutic clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of PEP (percent of patients using videos/complete questionnaires) | 3 years
  To assess the feasibility of implementing a PEP in the outpatient gastrointestinal malignancies service, at Sheba Medical Center, for patients undergoing active chemotherapy treatment. This outcome will be measured as percent of patients using the videos and percent of patients that complete the questionnaires.

SECONDARY OUTCOMES:
Secondary clinical outcomes 1 (mean number of referrals) | 3 years
  To monitor mean number of referrals to emergency room and admissions to the inpatient department.
Secondary clinical outcomes 2 (level of chemotoxicity) | 3 years
  To measure level of chemotoxicity - Neuropathy, diarrhea, nausea and vomiting, stomatitis and fever; using total number and percent of patients with side effects in each arm and Common Terminology Criteria for side effects (CTCAE) grading scale.
Secondary clinical outcomes 3 (Quality of Life) | 3 years
  To measure patient assessment of Quality of Life (QoL) using a validated questionnaire (QLQ-C30).
Secondary clinical outcomes 4 (treatment intensity and continuity) | 3 years
  To evaluate treatment intensity and continuity measured as number of chemotherapy cycles and cumulative chemotherapy dose.

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Margali, MD PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel